CLINICAL TRIAL: NCT03106922
Title: A Randomised, Single-blind, Active Controlled, Multi-centre Trial to Evaluate the Efficacy, Safety, Tolerability, Acceptability and Palatability of PMF104 Compared to a Conventional PEG-electrolyte Solution in Children Aged From 2 to Less Than 6, From 6 to Less Than 12, and Adolescents From 12 to Less Than 18 Years of Age Requiring a Diagnostic Procedure Concerning the Colon
Brief Title: A Trial to Evaluate the Efficacy and Safety of PMF104 Compared to a Conventional PEG-electrolyte Solution in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alfasigma S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PMF104 PD1-2-3/2013
Record Dates: First submitted 2017-03-27; First posted 2017-04-11 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2017-04

CONDITIONS: Bowel Preparation Before Colonoscopy
Keywords: Polyethylene glycol; Bowel cleansing; Colonoscopy
MeSH Terms: interventions — klean prep

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: During the study a single-blind design with respect to the investigational products will be achieved by providing the randomisation list only to the unblinded study staff personnel who will handle study drug management, preparation, dispensation and collection but who will not be involved in colonoscopy performing. The colonoscopy will be performed by experienced endoscopists who are unaware of the treatment actually being dispensed in each case. The endoscopist will be blinded by instructing all the other involved clinical staff, patients and patients' families to not discuss with him the specifics of the preparation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- PMF104 (Experimental): The day before the colonoscopy, starting in the mid-late afternoon (4-6 p.m.), by oral route:
  2<=Age<6
  * 500 ml in 1-1.5 hours <= to 18 kg
  * 625 ml in 1-1.5 hours >18 kg 6<=Age<12:
  * 750 ml in 1-2 hours <=25 kg
  * 1000 ml in 1-2 hours 25-35 kg
  * 1250 ml in 1-2 hours >35 kg 12>=Age<18 :
  * 1500 ml in 2-3 hours <= 45 kg
  * 1750 ml in 2-3 hours>45 kg.
  Rescue dose (if no clear watery stools 3 hours after the entire solution):
  * 250 ml 2 Age <=6;
  * 500 ml 6 <=Age<12; up to a cumulative maximum volume of 2000 ml 12<=Age<18.
  Interventions: Drug: PMF104
- Klean- prep (Active Comparator): The day before the colonoscopy, starting in the mid-late afternoon (4-6 p.m.), by oral route:
  * 2<=Age<6:
    * 90 ml/kg in 1-1.5 hours 2<=Age<6
    * 80 ml/kg in 1-1.5 hours 5<=Age<6
  * 2<=Age<6:
    * 80 ml/kg in 1-2 hours 6<=Age<10
    * 70 ml/kg in 1-2 hours 10<=Age<12
  * 12<=Age<18:
    * 70 ml/kg in 2-3 hours. Rescue dose (if no clear watery stools 3 hours after the entire Klean-Prep solution): 50% of the initial dose.
  Interventions: Drug: Klean-prep

INTERVENTIONS:
Drug: PMF104 — Powder for oral solution:
  * Sachet A: macrogol 4000 52.500 g, anhydrous sodium sulphate 3.750 g, simeticone 0.080 g;
  * Sachet B: sodium citrate 1.863 g, anhydrous citric acid 0.813 g, sodium chloride 0.730 g, potassium chloride 0.370 g;
  One sachet A + 1 sachet B in 500 ml of water
  Arms: PMF104
Drug: Klean-prep — Powder for oral solution:
  macrogol 3350 59.000 g, anhydrous sodium sulphate 5.685 g, sodium bicarbonate 1.685 g, sodium chloride 1.465 g, potassium chloride 0.7425 g.
  One sachet to be dissolved in 1 L of water
  Arms: Klean- prep

SUMMARY:
A randomised, single-blind, active controlled, multi-centre trial to evaluate the efficacy, safety, tolerability, acceptability and palatability of PMF104 compared to a conventional PEG-electrolyte solution in paediatric subjects requiring a diagnostic procedure concerning the colon.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the efficacy, safety, tolerability, acceptability and palatability of PMF104 compared to Klean-prep® in children aged from 2 to less than 18 years old requiring a diagnostic procedure of the colon.

Patients will be stratified according the following age strata:

* Children from 2 to less than 6 years of age (PMF104 PD1/13)
* Children from 6 to less than 12 years of age (PMF104 PD2/13)
* Children from 12 to less than 18 years of age (PMF104 PD3/13) The study will consist of a Screening Visit (V1), a Randomisation Visit (V2), a Drug Administration (Day 1), a Diagnostic Procedure (i.e. colonoscopy; V3) and a Follow-up Telephone Contact (FU).

At Screening Visit (V1) children will be evaluated for study eligibility, up to 11 days before the colonoscopy.

At Randomisation Visit (V2), if eligible, they will be randomised according to a single blind randomisation schedule in a 1:1 ratio to PMF104 or Klean-prep®; they will also receive the instructions to be followed for bowel preparation, and the questionnaire to be answered on the day of the bowel preparation. In case the Investigator will consider it as appropriate, the child will be hospitalised in the clinical facility the day before the colonoscopy in order to perform bowel preparation.

The day before the colonoscopy study drug will be administered orally starting in the mid-late afternoon (4-6 p.m.), as single dose.

The day of colonoscopy the diagnostic procedure will be performed blindly by an endoscopist unaware of the treatment administered to the subject, and both primary and secondary endpoints will be assessed.

On day 31 ± 2 (i.e. 30 ± 2 days after the day of the bowel preparation intake), the subjects will be contacted by a telephone call, to inquire about possible adverse events occurred after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged from 2 to less than 18 years during the entire study period undergoing elective colonoscopy;
2. Female subjects currently either of:

   * Non-childbearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is surgically sterilised via documented hysterectomy or bilateral tubal ligation), or
   * Childbearing potential: the subject is eligible to enter and participate in this study if she is not lactating and has a negative pregnancy test, and agrees to abstain from intercourses until the colonoscopy is performed (only menstruated females);
3. Patients whose parents/legal representatives have been thoroughly informed of the aim of the study procedures and provided signed and dated written informed consent;
4. Children aged from 6 to less than 12 years providing informed assent whenever possible;
5. Adolescents aged from 12 to less than 18 years providing informed assent;
6. Ability of the subjects and/or their parents/legal representatives to understand and comply with protocol requirements, instructions and protocol-stated restrictions.

Exclusion Criteria:

1. Requirement for urgent colonoscopy;
2. Gastrointestinal obstruction or perforation;
3. Bowel pseudo-obstruction;
4. Gastric retention;
5. Toxic colitis;
6. Toxic megacolon;
7. Known or suspected hypersensitivity to the active or other ingredients of both test product and reference product;
8. Clinically significant electrolyte imbalance;
9. Prior intestinal resection;
10. Structural abnormality of the lower gastrointestinal (GI) tract;
11. Known metabolic (particularly phenylketonuria), hepatic, renal or cardiac disease;
12. Congestive heart failure (NYHA class III and IV);
13. Known pregnancy;
14. Subject who have participated in another clinical trial or have taken an investigational drug within the last 3 months prior screening.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Estimated)
Dates: Start 2016-04; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Colon cleansing efficacy | Visit 3 (Day 2)
  Boston Bowel Preparation Scale score assessed blindly by the endoscopist

SECONDARY OUTCOMES:
Time to reach clear watery stools | Day 1
  The time when clear watery stools are obtained after completing the bowel solution
Proportion of patients in whom caecal intubation was achieved during colonoscopy | Visit 3 (Day 2)
  Proportion of patients in whom caecal intubation was achieved during colonoscopy
Proportion of patients achieving a BBPS score greater than or equal to 5 | Visit 3 (Day 2)
  Based on the BBPS score assigned during colonoscopy, each patient will be classified as being a "success" (patient achieving a BBPS score ≥ 5) or a "failure" (patient achieving a BBPS score < 5).
Proportion of patients that needs a rescue dose | Day 1
  Additional amount of test or reference will be given if patient will not have clear watery stools 3 hours after the administration of the scheduled amount of bowel solution
Compliance | Day 1
  Poor: intake of < 75% of the solution; Good: intake of at least 75% of the solution but <100%; Optimal: intake of the whole solution.
Acceptability | Day 1
  Pre-determined answers to question:"How difficult was to drink the bowel preparation solution?" 1 =Very difficult; 2 =Moderately difficult; 3 = Slightly difficult; 4 =Not difficult at all
Palatability | Day 1
  Pre-determined answers to question:"How did the solution taste?" 1 =Very bad; 2 = Bad; 3 =Good; 4 = Very good
Number of adverse events | From Visit 1 to Follow-up telephone contact
  Number of adverse events coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA).
Subjects withdrawn due to treatment emergent adverse events (TEAEs) | From Visit 1 to Follow-up telephone contact
  Number and percentage of patients withdrawn due to TEAEs
Tolerability Assessment | Visit 3 (Day 2)
  Recording of occurence and severity of nausea, vomiting, bloating, abdominal pain/cramps, anal irritation and fatigue/weakness, according to a 4 point scale:
  0 =No distress
  1. =Mild distress
  2. =Moderate distress
  3. = Severe distress

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Cucchiara, MD, Principal Investigator — Azienda Policlinico Umberto I
Locations (9):
- Pediatric Gastroenterology, Hepatology and Nutrition Children's University Hospital, Brussels, Belgium
- France (3):
  - Hôpital Jeanne de Flandre, Lille
  - University and Pediatric Hospital of Lyon, Lyon
  - Hôpital Armand-Trousseau, Paris
- Italy (5):
  - Ospedale Maggiore "C.A. Pizzardi" AUSL Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Meyer, Florence
  - Azienda Ospedaliera Universitaria "G. Martino", Messina
  - Azienda Policlinico Umberto I, Rome
  - Ospedale Pediatrico Bambino Gesù, Rome

IPD SHARING:
Plan to Share IPD: No